CLINICAL TRIAL: NCT02484391
Title: An Open Label Study to Evaluate the Feasibility of CPI-613 Given With High Dose Cytarabine and Mitoxantrone in Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: CPI-613, Cytarabine, and Mitoxantrone Hydrochloride in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia or Granulocytic Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00033779; NCI-2015-01002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00033779; CCCWFU 22215 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Granulocytic Sarcoma; Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Sarcoma, Myeloid; Leukemia, Myeloid, Acute | interventions — devimistat; Cytarabine; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613, cytarabine, mitoxantrone hydrochloride) (Experimental): See Detailed Description
  Interventions: Drug: 6,8-Bis(benzylthio)octanoic Acid; Drug: Cytarabine; Procedure: Hematopoietic Cell Transplantation; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: 6,8-Bis(benzylthio)octanoic Acid — Given IV
  Other Names: Alpha-Lipoic Acid Analogue CPI-613; CPI 613; CPI-613
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Hematopoietic Cell Transplantation — Undergo stem cell transplant
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This pilot phase I trial studies how well CPI-613 (6,8-bis[benzylthio]octanoic acid), cytarabine, and mitoxantrone hydrochloride work in treating patients with acute myeloid leukemia or granulocytic sarcoma (a malignant, green-colored tumor of myeloid cells [a type of immature white blood cell]) that has returned (relapsed) or that does not respond to treatment (refractory). 6,8-bis(benzylthio)octanoic acid is thought to kill cancer cells by turning off their mitochondria. Mitochondria are used by cancer cells to produce energy and are the building blocks needed to make more cancer cells. By shutting off these mitochondria, 6,8-bis(benzylthio)octanoic acid deprives the cancer cells of energy and other supplies that they need to survive and grow in the body. Drugs used in chemotherapy, such as cytarabine and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving 6,8-bis(benzylthio)octanoic acid together with cytarabine and mitoxantrone hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of CPI-613 when administered with high dose cytarabine, and mitoxantrone (mitoxantrone hydrochloride) in all three phases of salvage therapy (induction, consolidation and maintenance).

SECONDARY OBJECTIVES:

I. To observe the response rate (complete remission [CR], and CR with incomplete recovery [CRi]) of CPI-613 in combination with high dose cytarabine and mitoxantrone.

II. To observe the overall survival of patients treated with CPI-613 in combination with high dose cytarabine and mitoxantrone in induction, consolidation and maintenance.

III. To monitor toxicities experienced by patients treated with CPI-613 in combination with high dose cytarabine and mitoxantrone in induction, consolidation and maintenance.

OUTLINE:

SALVAGE INDUCTION COURSE 1: Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-5, cytarabine IV over 3 hours every 12 hours starting on day 3 for 5 doses, and mitoxantrone hydrochloride IV over 15 minutes after the first, third, and fifth doses of cytarabine.

SALVAGE INDUCTION COURSE 2 (OPTIONAL, AT DISCRETION OF TREATING PHYSICIAN): Patients receive 6,8-bis(benzylthio)octanoic acid, cytarabine, and mitoxantrone hydrochloride as in course 1 or an abbreviated second course at the discretion of the treating physician. In the abbreviated course, patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-3, cytarabine IV over 3 hours every 12 hours starting on day 2 for 3 doses, and mitoxantrone hydrochloride IV over 15 minutes after the first and third cytarabine doses.

SALVAGE CONSOLIDATION: Patients achieving response receive up to 2 courses of the abbreviated course of 6,8-bis(benzylthio)octanoic acid, high dose cytarabine, and mitoxantrone hydrochloride. Patients achieving response may undergo stem cell transplant at the discretion of the treating physician. Patients may proceed to maintenance after 1, 2 or no courses of consolidation at the discretion of the treating physician.

MAINTENANCE THERAPY: Patients achieving response receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented relapsed and/or refractory acute myeloid leukemia or granulocytic sarcoma
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists
* Mentally competent, ability to understand and willingness to sign the informed consent form
* No radiotherapy, treatment with cytotoxic agents (except CPI-613), treatment with biologic agents or any anti-cancer therapy within the 2 weeks prior to treatment with CPI-613; hydroxyurea and oral tyrosine kinase inhibitors being used without grade =< 2 toxicity can be taken until day 1 of therapy; patients must have fully recovered from the acute, non-hematological, non-infectious toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment); patients with persisting, non-hematologic, non-infectious toxicities from prior treatment =< grade 2 are eligible, but must be documented as such
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT)/serum glutamate pyruvate transaminase (SGPT) =< 3 x UNL (=< 5 x upper limit of normal [ULN] if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 umol/L
* International normalized ratio or INR must be < 1.5
* Left ventricular ejection fraction (by transthoracic echocardiography [TTE], multigated acquisition scan [MUGA] or cardiac magnetic resonance imaging [MRI]) sufficient to safely administer mitoxantrone as determined by the treating physician

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (e.g. symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, pericardial disease or New York Heart Association class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity
* Patients with active central nervous system (CNS) or epidural tumor
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 3 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Patients with large and recurrent pleural or peritoneal effusions requiring frequent drainage (e.g. weekly); patients with any amount of clinically significant pericardial effusion
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, uncontrolled arrhythmias, or symptomatic congestive heart failure
* Evidence of ongoing, uncontrolled infection
* Patients with known human immunodeficiency virus (HIV) infection
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 2 weeks prior to initiation of CPI-613 treatment (the use of Hydrea is allowed)
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* A history of additional risk factors for torsade de pointes (e.g., clinically significant heart failure, hypokalemia, family history of long QT syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayard Powell, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Anderson R, Miller LD, Isom S, Chou JW, Pladna KM, Schramm NJ, Ellis LR, Howard DS, Bhave RR, Manuel M, Dralle S, Lyerly S, Powell BL, Pardee TS. Phase II trial of cytarabine and mitoxantrone with devimistat in acute myeloid leukemia. Nat Commun. 2022 Mar 30;13(1):1673. doi: 10.1038/s41467-022-29039-4. PMID 35354808

RESULTS

PARTICIPANT FLOW:
Groups:
- 1500: 1500 mg/m2 devimistat
- 2000: 2000 mg/m2 devimistat
- 2500: 2500 mg/m2 devimistat
Period: Overall Study
Arm/Group | 1500 | 2000 | 2500
Started | 21 | 20 | 7
Achieved Remission | 9 | 7 | 5
Received Maintenance Therapy | 0 | 0 | 2
Completed | 0 | 0 | 0
Not Completed | 21 | 20 | 7
Not completed — Lack of Efficacy | 15 | 14 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Physician Decision | 1 | 3 | 0
Not completed — Went to Transplant | 5 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1500 | 2000 | 2500 | Total
Number analyzed (Participants) | 21 | 20 | 7 | 48
Age, Continuous [Median (Full Range); unit: years] | 61 [35 to 85] | 65.5 [21 to 76] | 64 [27 to 78] | 64 [21 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 3 | 20
  Male | 12 | 12 | 4 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 1 | 7
  White | 18 | 16 | 6 | 40
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Administering CPI-613 in Combination With High Dose Cytarabine and Mitoxantrone During Induction, Consolidation and Maintenance Therapies, Defined as Percentage of Patients Eligible for Maintenance Therapy Who Complete at Least 3 Courses
Description: Feasibility is determined by the percentage of patients eligible for maintenance therapy who complete at least 3 cycles, if ≥50% of eligible patients complete 3 cycles of maintenance therapy we will consider this regimen feasible for future study.
Time Frame: Up to 12 weeks of maintenance therapy
Population: None of the 9 participants in the 1500 mg arm and the 7 participants in the 2000 mg arm started maintenance, only 2 out of the 5 participants in the 2500 mg arm started maintenance. None of participants completed three cycles of maintenance.
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 0 | 0 | 2
Participants
  Started maintenance therapy | 0 | 0 | 2
  Completed 3 cycles of maintenance therapy | 0 | 0 | 0

2. Secondary Outcome: Frequency of Toxicities Experienced by the Participants, Graded Using the National Cancer Institute Common Terminology Criteria for Adverse Events 3.0
Description: The frequency of toxicities experienced by the participants will be presented by type and grade in an effort to monitor and report safety of the treatment. Showing grade 2 and greater event and the highest grade of each type per participant so that a participant is only evaluated once per toxicity type. Reporting events where at least 10% (n=5) of study participants reported a grade 2 or greater event.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 21 | 20 | 7
Participants
  Abdominal pain: Grade 2 | 3 | 1 | 5
  Abdominal pain: Grade 3 | 0 | 1 | 1
  Abdominal pain: Grade 4 | 0 | 0 | 0
  Abdominal pain: Grade 5 | 0 | 0 | 0
  Abdominal pain: Not observed or Grade 1 | 18 | 18 | 1
  Activated partial thromboplastin time prolonged: Grade 2 | 2 | 0 | 1
  Activated partial thromboplastin time prolonged: Grade 3 | 2 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 4 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Grade 5 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged: Not observed or Grade 1 | 17 | 20 | 6
  Acute kidney injury: Grade 2 | 2 | 1 | 0
  Acute kidney injury: Grade 3 | 0 | 0 | 1
  Acute kidney injury: Grade 4 | 3 | 0 | 0
  Acute kidney injury: Grade 5 | 0 | 0 | 0
  Acute kidney injury: Not observed or Grade 1 | 16 | 19 | 6
  Agitation: Grade 2 | 2 | 1 | 0
  Agitation: Grade 3 | 2 | 0 | 0
  Agitation: Grade 4 | 0 | 0 | 0
  Agitation: Grade 5 | 0 | 0 | 0
  Agitation: Not observed or Grade 1 | 17 | 19 | 7
  Alanine aminotransferase increased: Grade 2 | 3 | 2 | 1
  Alanine aminotransferase increased: Grade 3 | 1 | 1 | 1
  Alanine aminotransferase increased: Grade 4 | 0 | 0 | 0
  Alanine aminotransferase increased: Grade 5 | 0 | 0 | 0
  Alanine aminotransferase increased: Not observed or Grade 1 | 17 | 17 | 5
  Alkalosis: Grade 2 | 0 | 0 | 0
  Alkalosis: Grade 3 | 2 | 3 | 0
  Alkalosis: Grade 4 | 0 | 0 | 0
  Alkalosis: Grade 5 | 0 | 0 | 0
  Alkalosis: Not observed or Grade 1 | 19 | 17 | 7
  Anemia: Grade 2 | 1 | 0 | 0
  Anemia: Grade 3 | 19 | 19 | 6
  Anemia: Grade 4 | 1 | 0 | 1
  Anemia: Grade 5 | 0 | 0 | 0
  Anemia: Not observed or Grade 1 | 0 | 1 | 0
  Anorexia: Grade 2 | 9 | 8 | 4
  Anorexia: Grade 3 | 4 | 8 | 2
  Anorexia: Grade 4 | 0 | 0 | 0
  Anorexia: Grade 5 | 0 | 0 | 0
  Anorexia: Not observed or Grade 1 | 8 | 4 | 1
  Anxiety: Grade 2 | 5 | 7 | 5
  Anxiety: Grade 3 | 0 | 0 | 0
  Anxiety: Grade 4 | 0 | 0 | 0
  Anxiety: Grade 5 | 0 | 0 | 0
  Anxiety: Not observed or Grade 1 | 16 | 13 | 2
  Aspartate aminotransferase increased: Grade 2 | 2 | 3 | 1
  Aspartate aminotransferase increased: Grade 3 | 3 | 1 | 1
  Aspartate aminotransferase increased: Grade 4 | 0 | 0 | 0
  Aspartate aminotransferase increased: Grade 5 | 0 | 0 | 0
  Aspartate aminotransferase increased: Not observed or Grade 1 | 16 | 16 | 5
  Back pain: Grade 2 | 2 | 5 | 4
  Back pain: Grade 3 | 0 | 0 | 0
  Back pain: Grade 4 | 0 | 0 | 0
  Back pain: Grade 5 | 0 | 0 | 0
  Back pain: Not observed or Grade 1 | 19 | 15 | 3
  Blood and lymphatic system disorders - Other: Grade 2 | 4 | 1 | 0
  Blood and lymphatic system disorders - Other: Grade 3 | 0 | 0 | 0
  Blood and lymphatic system disorders - Other: Grade 4 | 0 | 0 | 0
  Blood and lymphatic system disorders - Other: Grade 5 | 0 | 0 | 0
  Blood and lymphatic system disorders - Other: Not observed or Grade 1 | 17 | 19 | 7
  Blood bilirubin increased: Grade 2 | 5 | 5 | 2
  Blood bilirubin increased: Grade 3 | 2 | 5 | 0
  Blood bilirubin increased: Grade 4 | 0 | 0 | 0
  Blood bilirubin increased: Grade 5 | 0 | 0 | 0
  Blood bilirubin increased: Not observed or Grade 1 | 14 | 10 | 5
  Cardiac troponin I increased: Grade 2 | 0 | 0 | 0
  Cardiac troponin I increased: Grade 3 | 3 | 2 | 0
  Cardiac troponin I increased: Grade 4 | 0 | 0 | 0
  Cardiac troponin I increased: Grade 5 | 0 | 0 | 0
  Cardiac troponin I increased: Not observed or Grade 1 | 18 | 18 | 7
  Catheter related infection: Grade 2 | 0 | 0 | 0
  Catheter related infection: Grade 3 | 2 | 6 | 0
  Catheter related infection: Grade 4 | 1 | 1 | 0
  Catheter related infection: Grade 5 | 0 | 0 | 0
  Catheter related infection: Not observed or Grade 1 | 18 | 13 | 7
  Chills: Grade 2 | 2 | 1 | 0
  Chills: Grade 3 | 1 | 1 | 0
  Chills: Grade 4 | 0 | 0 | 0
  Chills: Grade 5 | 0 | 0 | 0
  Chills: Not observed or Grade 1 | 18 | 18 | 7
  Chronic kidney disease: Grade 2 | 3 | 11 | 2
  Chronic kidney disease: Grade 3 | 1 | 0 | 0
  Chronic kidney disease: Grade 4 | 2 | 0 | 1
  Chronic kidney disease: Grade 5 | 0 | 0 | 0
  Chronic kidney disease: Not observed or Grade 1 | 15 | 9 | 4
  Confusion: Grade 2 | 4 | 2 | 2
  Confusion: Grade 3 | 0 | 0 | 0
  Confusion: Grade 4 | 0 | 0 | 0
  Confusion: Grade 5 | 0 | 0 | 0
  Confusion: Not observed or Grade 1 | 17 | 18 | 5
  Creatinine increased: Grade 2 | 2 | 0 | 0
  Creatinine increased: Grade 3 | 3 | 0 | 1
  Creatinine increased: Grade 4 | 0 | 0 | 0
  Creatinine increased: Grade 5 | 0 | 0 | 0
  Creatinine increased: Not observed or Grade 1 | 16 | 20 | 6
  Dehydration: Grade 2 | 1 | 1 | 2
  Dehydration: Grade 3 | 0 | 0 | 1
  Dehydration: Grade 4 | 0 | 0 | 0
  Dehydration: Grade 5 | 0 | 0 | 0
  Dehydration: Not observed or Grade 1 | 20 | 19 | 4
  Delirium: Grade 2 | 4 | 1 | 0
  Delirium: Grade 3 | 2 | 0 | 0
  Delirium: Grade 4 | 0 | 0 | 0
  Delirium: Grade 5 | 0 | 0 | 0
  Delirium: Not observed or Grade 1 | 15 | 19 | 7
  Depression: Grade 2 | 2 | 3 | 2
  Depression: Grade 3 | 0 | 0 | 0
  Depression: Grade 4 | 0 | 0 | 0
  Depression: Grade 5 | 0 | 0 | 0
  Depression: Not observed or Grade 1 | 19 | 17 | 5
  Diarrhea: Grade 2 | 5 | 9 | 2
  Diarrhea: Grade 3 | 5 | 6 | 4
  Diarrhea: Grade 4 | 0 | 0 | 0
  Diarrhea: Grade 5 | 0 | 0 | 0
  Diarrhea: Not observed or Grade 1 | 11 | 5 | 1
  Disseminated intravascular coagulation: Grade 2 | 14 | 18 | 7
  Disseminated intravascular coagulation: Grade 3 | 1 | 0 | 0
  Disseminated intravascular coagulation: Grade 4 | 0 | 0 | 0
  Disseminated intravascular coagulation: Grade 5 | 0 | 0 | 0
  Disseminated intravascular coagulation: Not observed or Grade 1 | 6 | 2 | 0
  Dysgeusia: Grade 2 | 1 | 4 | 0
  Dysgeusia: Grade 3 | 0 | 0 | 0
  Dysgeusia: Grade 4 | 0 | 0 | 0
  Dysgeusia: Grade 5 | 0 | 0 | 0
  Dysgeusia: Not observed or Grade 1 | 20 | 16 | 7
  Dysphagia: Grade 2 | 5 | 1 | 0
  Dysphagia: Grade 3 | 2 | 1 | 1
  Dysphagia: Grade 4 | 0 | 0 | 0
  Dysphagia: Grade 5 | 0 | 0 | 0
  Dysphagia: Not observed or Grade 1 | 14 | 18 | 6
  Dyspnea: Grade 2 | 3 | 6 | 0
  Dyspnea: Grade 3 | 2 | 4 | 1
  Dyspnea: Grade 4 | 1 | 1 | 0
  Dyspnea: Grade 5 | 0 | 0 | 0
  Dyspnea: Not observed or Grade 1 | 15 | 9 | 6
  Edema limbs: Grade 2 | 4 | 2 | 0
  Edema limbs: Grade 3 | 0 | 0 | 1
  Edema limbs: Grade 4 | 0 | 0 | 0
  Edema limbs: Grade 5 | 0 | 0 | 0
  Edema limbs: Not observed or Grade 1 | 17 | 18 | 6
  Ejection fraction decreased: Grade 2 | 2 | 5 | 1
  Ejection fraction decreased: Grade 3 | 1 | 0 | 0
  Ejection fraction decreased: Grade 4 | 0 | 0 | 0
  Ejection fraction decreased: Grade 5 | 0 | 0 | 0
  Ejection fraction decreased: Not observed or Grade 1 | 18 | 15 | 6
  Electrocardiogram QT corrected interval prolonged: Grade 2 | 2 | 4 | 4
  Electrocardiogram QT corrected interval prolonged: Grade 3 | 0 | 1 | 0
  Electrocardiogram QT corrected interval prolonged: Grade 4 | 0 | 0 | 0
  Electrocardiogram QT corrected interval prolonged: Grade 5 | 0 | 0 | 0
  Electrocardiogram QT corrected interval prolonged: Not observed or Grade 1 | 19 | 15 | 3
  Epistaxis: Grade 2 | 1 | 1 | 0
  Epistaxis: Grade 3 | 2 | 1 | 1
  Epistaxis: Grade 4 | 0 | 0 | 0
  Epistaxis: Grade 5 | 0 | 0 | 0
  Epistaxis: Not observed or Grade 1 | 18 | 18 | 6
  Fatigue: Grade 2 | 8 | 10 | 3
  Fatigue: Grade 3 | 2 | 4 | 3
  Fatigue: Grade 4 | 0 | 0 | 0
  Fatigue: Grade 5 | 0 | 0 | 0
  Fatigue: Not observed or Grade 1 | 11 | 6 | 1
  Febrile neutropenia: Grade 2 | 0 | 0 | 0
  Febrile neutropenia: Grade 3 | 6 | 13 | 4
  Febrile neutropenia: Grade 4 | 0 | 1 | 0
  Febrile neutropenia: Grade 5 | 0 | 0 | 0
  Febrile neutropenia: Not observed or Grade 1 | 15 | 6 | 3
  Fever: Grade 2 | 12 | 9 | 3
  Fever: Grade 3 | 0 | 3 | 0
  Fever: Grade 4 | 0 | 0 | 0
  Fever: Grade 5 | 0 | 0 | 0
  Fever: Not observed or Grade 1 | 9 | 8 | 4
  Gastrointestinal disorders - Other: Grade 2 | 1 | 3 | 5
  Gastrointestinal disorders - Other: Grade 3 | 0 | 2 | 0
  Gastrointestinal disorders - Other: Grade 4 | 0 | 1 | 0
  Gastrointestinal disorders - Other: Grade 5 | 0 | 0 | 0
  Gastrointestinal disorders - Other: Not observed or Grade 1 | 20 | 14 | 2
  Generalized muscle weakness: Grade 2 | 4 | 2 | 3
  Generalized muscle weakness: Grade 3 | 2 | 5 | 1
  Generalized muscle weakness: Grade 4 | 0 | 0 | 0
  Generalized muscle weakness: Grade 5 | 0 | 0 | 0
  Generalized muscle weakness: Not observed or Grade 1 | 15 | 13 | 3
  Headache: Grade 2 | 3 | 4 | 1
  Headache: Grade 3 | 2 | 2 | 3
  Headache: Grade 4 | 0 | 0 | 0
  Headache: Grade 5 | 0 | 0 | 0
  Headache: Not observed or Grade 1 | 16 | 14 | 3
  Hyperglycemia: Grade 2 | 6 | 6 | 0
  Hyperglycemia: Grade 3 | 5 | 3 | 2
  Hyperglycemia: Grade 4 | 0 | 0 | 0
  Hyperglycemia: Grade 5 | 0 | 0 | 0
  Hyperglycemia: Not observed or Grade 1 | 10 | 11 | 5
  Hypertension: Grade 2 | 3 | 2 | 2
  Hypertension: Grade 3 | 5 | 3 | 0
  Hypertension: Grade 4 | 0 | 0 | 0
  Hypertension: Grade 5 | 0 | 0 | 0
  Hypertension: Not observed or Grade 1 | 13 | 15 | 5
  Hypoalbuminemia: Grade 2 | 13 | 16 | 3
  Hypoalbuminemia: Grade 3 | 1 | 0 | 1
  Hypoalbuminemia: Grade 4 | 3 | 0 | 0
  Hypoalbuminemia: Grade 5 | 0 | 0 | 0
  Hypoalbuminemia: Not observed or Grade 1 | 4 | 4 | 3
  Hypocalcemia: Grade 2 | 1 | 9 | 3
  Hypocalcemia: Grade 3 | 3 | 1 | 1
  Hypocalcemia: Grade 4 | 2 | 0 | 0
  Hypocalcemia: Grade 5 | 0 | 0 | 0
  Hypocalcemia: Not observed or Grade 1 | 15 | 10 | 3
  Hypokalemia: Grade 2 | 2 | 1 | 0
  Hypokalemia: Grade 3 | 7 | 8 | 3
  Hypokalemia: Grade 4 | 0 | 2 | 0
  Hypokalemia: Grade 5 | 0 | 0 | 0
  Hypokalemia: Not observed or Grade 1 | 12 | 9 | 4
  Hypomagnesemia: Grade 2 | 4 | 1 | 2
  Hypomagnesemia: Grade 3 | 0 | 0 | 0
  Hypomagnesemia: Grade 4 | 0 | 0 | 0
  Hypomagnesemia: Grade 5 | 0 | 0 | 0
  Hypomagnesemia: Not observed or Grade 1 | 17 | 19 | 5
  Hyponatremia: Grade 2 | 1 | 0 | 0
  Hyponatremia: Grade 3 | 1 | 0 | 1
  Hyponatremia: Grade 4 | 3 | 0 | 0
  Hyponatremia: Grade 5 | 0 | 0 | 0
  Hyponatremia: Not observed or Grade 1 | 16 | 20 | 6
  Hypophosphatemia: Grade 2 | 7 | 8 | 0
  Hypophosphatemia: Grade 3 | 6 | 6 | 6
  Hypophosphatemia: Grade 4 | 0 | 2 | 0
  Hypophosphatemia: Grade 5 | 0 | 0 | 0
  Hypophosphatemia: Not observed or Grade 1 | 8 | 4 | 1
  Hypotension: Grade 2 | 2 | 3 | 4
  Hypotension: Grade 3 | 2 | 2 | 0
  Hypotension: Grade 4 | 0 | 0 | 0
  Hypotension: Grade 5 | 0 | 0 | 0
  Hypotension: Not observed or Grade 1 | 17 | 15 | 3
  Hypoxia: Grade 2 | 0 | 1 | 0
  Hypoxia: Grade 3 | 2 | 3 | 1
  Hypoxia: Grade 4 | 1 | 1 | 0
  Hypoxia: Grade 5 | 0 | 0 | 0
  Hypoxia: Not observed or Grade 1 | 18 | 15 | 6
  Infections and infestations - Other: Grade 2 | 2 | 3 | 0
  Infections and infestations - Other: Grade 3 | 2 | 5 | 3
  Infections and infestations - Other: Grade 4 | 1 | 0 | 0
  Infections and infestations - Other: Grade 5 | 0 | 0 | 0
  Infections and infestations - Other: Not observed or Grade 1 | 16 | 12 | 4
  Insomnia: Grade 2 | 4 | 4 | 0
  Insomnia: Grade 3 | 0 | 0 | 0
  Insomnia: Grade 4 | 0 | 0 | 0
  Insomnia: Grade 5 | 0 | 0 | 0
  Insomnia: Not observed or Grade 1 | 17 | 16 | 7
  Lung infection: Grade 2 | 4 | 2 | 0
  Lung infection: Grade 3 | 1 | 9 | 2
  Lung infection: Grade 4 | 0 | 0 | 0
  Lung infection: Grade 5 | 1 | 0 | 0
  Lung infection: Not observed or Grade 1 | 15 | 9 | 5
  Lymphocyte count decreased: Grade 2 | 0 | 0 | 0
  Lymphocyte count decreased: Grade 3 | 0 | 1 | 0
  Lymphocyte count decreased: Grade 4 | 21 | 19 | 7
  Lymphocyte count decreased: Grade 5 | 0 | 0 | 0
  Lymphocyte count decreased: Not observed or Grade 1 | 0 | 0 | 0
  Mucositis oral: Grade 2 | 1 | 2 | 0
  Mucositis oral: Grade 3 | 0 | 2 | 1
  Mucositis oral: Grade 4 | 0 | 0 | 0
  Mucositis oral: Grade 5 | 0 | 0 | 0
  Mucositis oral: Not observed or Grade 1 | 20 | 16 | 6
  Nausea: Grade 2 | 6 | 8 | 4
  Nausea: Grade 3 | 0 | 5 | 3
  Nausea: Grade 4 | 0 | 0 | 0
  Nausea: Grade 5 | 0 | 0 | 0
  Nausea: Not observed or Grade 1 | 15 | 7 | 0
  Neck pain: Grade 2 | 2 | 0 | 1
  Neck pain: Grade 3 | 1 | 1 | 0
  Neck pain: Grade 4 | 0 | 0 | 0
  Neck pain: Grade 5 | 0 | 0 | 0
  Neck pain: Not observed or Grade 1 | 18 | 19 | 6
  Neutrophil count decreased: Grade 2 | 0 | 0 | 0
  Neutrophil count decreased: Grade 3 | 0 | 0 | 0
  Neutrophil count decreased: Grade 4 | 21 | 19 | 7
  Neutrophil count decreased: Grade 5 | 0 | 0 | 0
  Neutrophil count decreased: Not observed or Grade 1 | 0 | 1 | 0
  Non-cardiac chest pain: Grade 2 | 2 | 2 | 1
  Non-cardiac chest pain: Grade 3 | 1 | 1 | 0
  Non-cardiac chest pain: Grade 4 | 0 | 0 | 0
  Non-cardiac chest pain: Grade 5 | 0 | 0 | 0
  Non-cardiac chest pain: Not observed or Grade 1 | 18 | 17 | 6
  Oral pain: Grade 2 | 0 | 3 | 1
  Oral pain: Grade 3 | 0 | 1 | 0
  Oral pain: Grade 4 | 0 | 0 | 0
  Oral pain: Grade 5 | 0 | 0 | 0
  Oral pain: Not observed or Grade 1 | 21 | 16 | 6
  Pain: Grade 2 | 4 | 1 | 2
  Pain: Grade 3 | 1 | 1 | 3
  Pain: Grade 4 | 0 | 0 | 0
  Pain: Grade 5 | 0 | 0 | 0
  Pain: Not observed or Grade 1 | 16 | 18 | 2
  Pain in extremity: Grade 2 | 4 | 0 | 1
  Pain in extremity: Grade 3 | 0 | 1 | 3
  Pain in extremity: Grade 4 | 0 | 0 | 0
  Pain in extremity: Grade 5 | 0 | 0 | 0
  Pain in extremity: Not observed or Grade 1 | 17 | 19 | 3
  Platelet count decreased: Grade 2 | 0 | 0 | 0
  Platelet count decreased: Grade 3 | 0 | 0 | 0
  Platelet count decreased: Grade 4 | 21 | 20 | 7
  Platelet count decreased: Grade 5 | 0 | 0 | 0
  Platelet count decreased: Not observed or Grade 1 | 0 | 0 | 0
  Proteinuria: Grade 2 | 1 | 1 | 1
  Proteinuria: Grade 3 | 2 | 0 | 0
  Proteinuria: Grade 4 | 0 | 0 | 0
  Proteinuria: Grade 5 | 0 | 0 | 0
  Proteinuria: Not observed or Grade 1 | 18 | 19 | 6
  Pulmonary edema: Grade 2 | 2 | 1 | 0
  Pulmonary edema: Grade 3 | 1 | 1 | 0
  Pulmonary edema: Grade 4 | 0 | 0 | 0
  Pulmonary edema: Grade 5 | 0 | 0 | 0
  Pulmonary edema: Not observed or Grade 1 | 18 | 18 | 7
  Respiratory failure: Grade 2 | 0 | 0 | 0
  Respiratory failure: Grade 3 | 0 | 0 | 0
  Respiratory failure: Grade 4 | 5 | 2 | 0
  Respiratory failure: Grade 5 | 0 | 0 | 0
  Respiratory failure: Not observed or Grade 1 | 16 | 18 | 7
  Respiratory, thoracic and mediastinal disorders - Other: Grade 2 | 4 | 1 | 0
  Respiratory, thoracic and mediastinal disorders - Other: Grade 3 | 1 | 1 | 0
  Respiratory, thoracic and mediastinal disorders - Other: Grade 4 | 1 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Other: Grade 5 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders - Other: Not observed or Grade 1 | 15 | 18 | 7
  Sinus tachycardia: Grade 2 | 4 | 1 | 0
  Sinus tachycardia: Grade 3 | 1 | 0 | 0
  Sinus tachycardia: Grade 4 | 0 | 0 | 0
  Sinus tachycardia: Grade 5 | 0 | 0 | 0
  Sinus tachycardia: Not observed or Grade 1 | 16 | 19 | 7
  Sinusitis: Grade 2 | 2 | 0 | 0
  Sinusitis: Grade 3 | 1 | 0 | 1
  Sinusitis: Grade 4 | 0 | 1 | 0
  Sinusitis: Grade 5 | 0 | 0 | 0
  Sinusitis: Not observed or Grade 1 | 18 | 19 | 6
  Skin and subcutaneous tissue disorders - Other: Grade 2 | 1 | 3 | 1
  Skin and subcutaneous tissue disorders - Other: Grade 3 | 1 | 1 | 0
  Skin and subcutaneous tissue disorders - Other: Grade 4 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Other: Grade 5 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders - Other: Not observed or Grade 1 | 19 | 16 | 6
  Somnolence: Grade 2 | 1 | 1 | 1
  Somnolence: Grade 3 | 1 | 0 | 0
  Somnolence: Grade 4 | 0 | 0 | 0
  Somnolence: Grade 5 | 1 | 0 | 0
  Somnolence: Not observed or Grade 1 | 18 | 19 | 6
  Sore throat: Grade 2 | 2 | 0 | 0
  Sore throat: Grade 3 | 0 | 3 | 1
  Sore throat: Grade 4 | 0 | 0 | 0
  Sore throat: Grade 5 | 0 | 0 | 0
  Sore throat: Not observed or Grade 1 | 19 | 17 | 6
  Vomiting: Grade 2 | 1 | 3 | 2
  Vomiting: Grade 3 | 1 | 2 | 1
  Vomiting: Grade 4 | 0 | 0 | 0
  Vomiting: Grade 5 | 0 | 0 | 0
  Vomiting: Not observed or Grade 1 | 19 | 15 | 4
  Weight gain: Grade 2 | 4 | 2 | 2
  Weight gain: Grade 3 | 0 | 0 | 1
  Weight gain: Grade 4 | 0 | 0 | 0
  Weight gain: Grade 5 | 0 | 0 | 0
  Weight gain: Not observed or Grade 1 | 17 | 18 | 4
  Weight loss: Grade 2 | 0 | 9 | 2
  Weight loss: Grade 3 | 0 | 0 | 1
  Weight loss: Grade 4 | 0 | 0 | 0
  Weight loss: Grade 5 | 0 | 0 | 0
  Weight loss: Not observed or Grade 1 | 21 | 11 | 4
  White blood cell decreased: Grade 2 | 0 | 0 | 0
  White blood cell decreased: Grade 3 | 0 | 0 | 0
  White blood cell decreased: Grade 4 | 21 | 19 | 7
  White blood cell decreased: Grade 5 | 0 | 0 | 0
  White blood cell decreased: Not observed or Grade 1 | 0 | 1 | 0

3. Secondary Outcome: Overall Survival
Description: Will use Kaplan-Meier estimation to analyze overall survival.
Time Frame: Time from enrollment on trial to death from any cause, assessed up to 30 months after completion of therapy
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 21 | 20 | 7
months | 5.4 [1.7 to 7.8] | 7.8 [1.8 to 14.1] | 10 [3.0 to 12.5]

4. Secondary Outcome: Response Rate (CR and CRi), Assessed by Standard Criteria for AML
Description: Confidence intervals will be calculated around the estimates of the response rate (CR and CRi). Assuming a response rate of 0.5, with 50 participants, 95 percent confidence intervals can be created with a 0.14 margin of error (0.36, 0.64).
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 21 | 20 | 7
Participants | 9 | 7 | 5

5. Other Pre Specified Outcome: Early Mortality (Death Within 60 Days of Beginning of Treatment)
Description: Early mortality (death within 60 days of beginning of treatment).
Time Frame: Up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 21 | 20 | 7
Participants
  Alive at day 60 | 15 | 14 | 6
  Deceased at day 60 | 6 | 6 | 1

6. Other Pre Specified Outcome: Complete Response
Description: Complete response rates
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | 1500 | 2000 | 2500
Number analyzed (Participants) | 21 | 20 | 7
Participants | 8 | 5 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events were collected while patients were on treatment, which ranged from 15 days to 187 days (up to 6 months)
Description: Serious adverse events include all unexpected grade 4 and all grade 5 adverse events.
Arm/Group | 1500 | 2000 | 2500
All-Cause Mortality (participants affected / at risk) | 6/21 | 6/20 | 1/7
Serious Adverse Events (participants affected / at risk) | 21/21 | 16/20 | 4/7
Other Adverse Events (participants affected / at risk) | 21/21 | 20/20 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1500 (N=21) | 2000 (N=20) | 2500 (N=7)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 17 (27) | 3 (15) | 1 (5)
Neutrophil count decreased (Investigations) | 15 (24) | 2 (19) | 1 (5)
Platelet count decreased (Investigations) | 16 (31) | 3 (19) | 1 (6)
White blood cell decreased (Investigations) | 16 (27) | 2 (19) | 1 (5)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cardiac disorders - Other: (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other: (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other: (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other: (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other: (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1500 (N=21) | 2000 (N=20) | 2500 (N=7)
Anemia (Blood and lymphatic system disorders) | 20 (38) | 19 (36) | 6 (14)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 15 (21) | 18 (27) | 7 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 6 (8) | 13 (14) | 4 (4)
Blood and lymphatic system disorders - Other: (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 3 (3) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 8 (9) | 13 (14) | 4 (6)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac disorders - Other: (Cardiac disorders) | 2 (2) | 6 (7) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other: (Eye disorders) | 4 (4) | 3 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (10) | 5 (6) | 6 (8)
Anal pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (12) | 8 (9) | 4 (6)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 16 (22) | 20 (30) | 7 (11)
Dry mouth (Gastrointestinal disorders) | 9 (10) | 9 (10) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 4 (4) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (6) | 11 (13) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (22) | 16 (24) | 7 (11)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (13) | 10 (17) | 4 (7)
Gastrointestinal disorders - Other: (Gastrointestinal disorders) | 5 (5) | 9 (20) | 5 (8)
Chills (General disorders) | 11 (13) | 7 (8) | 4 (4)
Edema face (General disorders) | 3 (3) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 12 (13) | 14 (21) | 4 (7)
Edema trunk (General disorders) | 2 (2) | 0 (0) | 1 (1)
Facial pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 16 (25) | 17 (27) | 7 (10)
Fever (General disorders) | 15 (20) | 14 (17) | 6 (7)
Gait disturbance (General disorders) | 3 (3) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 3 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 7 (8) | 7 (9) | 4 (4)
Pain (General disorders) | 7 (9) | 11 (12) | 5 (9)
General disorders and administration site conditions - Other: (General disorders) | 2 (2) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 3 (3) | 6 (6) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 5 (5) | 11 (11) | 2 (3)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infections and infestations - Other: (Infections and infestations) | 4 (5) | 6 (10) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 4 (4) | 5 (7) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other: (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 8 (9) | 10 (13) | 6 (8)
Alanine aminotransferase increased (Investigations) | 16 (20) | 14 (19) | 7 (9)
Alkaline phosphatase increased (Investigations) | 10 (13) | 9 (12) | 4 (6)
Aspartate aminotransferase increased (Investigations) | 18 (22) | 15 (21) | 7 (9)
Blood bilirubin increased (Investigations) | 14 (16) | 15 (22) | 7 (8)
Cardiac troponin I increased (Investigations) | 3 (3) | 5 (6) | 0 (0)
Creatinine increased (Investigations) | 6 (6) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 3 (3) | 5 (6) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 3 (3) | 10 (12) | 4 (6)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (12) | 17 (22) | 6 (10)
Neutrophil count decreased (Investigations) | 6 (12) | 17 (17) | 6 (9)
Platelet count decreased (Investigations) | 5 (9) | 17 (18) | 6 (9)
Weight gain (Investigations) | 5 (6) | 7 (9) | 5 (6)
Weight loss (Investigations) | 4 (6) | 13 (20) | 4 (6)
White blood cell decreased (Investigations) | 5 (13) | 17 (17) | 6 (10)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 16 (23) | 17 (25) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (37) | 19 (36) | 7 (14)
Hypermagnesemia (Metabolism and nutrition disorders) | 6 (7) | 6 (6) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 (30) | 20 (34) | 7 (12)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (18) | 17 (20) | 6 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 18 (23) | 17 (27) | 7 (11)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (25) | 18 (30) | 6 (11)
Hyponatremia (Metabolism and nutrition disorders) | 10 (14) | 10 (12) | 6 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (16) | 15 (18) | 6 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (10) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (10) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 2 (2) | 6 (11)
Musculoskeletal and connective tissue disorder - Other: (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 6 (8) | 3 (3)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 9 (9) | 11 (15) | 2 (3)
Encephalopathy (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 9 (11) | 13 (16) | 5 (8)
Lethargy (Nervous system disorders) | 4 (4) | 2 (2) | 2 (2)
Movements involuntary (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 4 (4) | 6 (6) | 3 (3)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 3 (5) | 0 (0)
Nervous system disorders - Other: (Nervous system disorders) | 4 (8) | 2 (2) | 2 (3)
Agitation (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 8 (8) | 10 (12) | 5 (6)
Confusion (Psychiatric disorders) | 6 (6) | 7 (7) | 3 (4)
Delirium (Psychiatric disorders) | 6 (6) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 7 (9) | 3 (4) | 2 (3)
Hallucinations (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (7) | 6 (7) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 2 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 5 (6) | 11 (14) | 3 (5)
Hematuria (Renal and urinary disorders) | 6 (6) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (4) | 5 (5) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 5 (5) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 5 (5) | 1 (1)
Renal and urinary disorders - Other: (Renal and urinary disorders) | 3 (6) | 2 (3) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other: (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (9) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (18) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 7 (7) | 3 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (9) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other: (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (9) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7) | 9 (11) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (12) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6) | 1 (1)
Skin and subcutaneous tissue disorders - Other: (Skin and subcutaneous tissue disorders) | 4 (8) | 12 (22) | 6 (10)
Hot flashes (Vascular disorders) | 6 (6) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 5 (6) | 2 (2)
Hypotension (Vascular disorders) | 5 (6) | 5 (7) | 4 (6)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT02484391/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT02484391/ICF_000.pdf